CLINICAL TRIAL: NCT02740114
Title: Wound Infiltration With Liposomal Bupivacaine vs. Standard Wound Infiltration With Bupivacaine in Patient's Undergoing Open Gynecologic Surgery on an Enhanced Recovery Pathway: A Single-Blinded, Randomized, Controlled Study
Brief Title: Wound Infiltration With Liposomal Bupivacaine vs. Standard Wound Infiltration With Bupivacaine in Patient's Undergoing Open Gynecologic Surgery on an Enhanced Recovery Pathway
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per PIs request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-1119; NCI-2016-00739 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Malignant Neoplasms of Female Genital Organs; Gynecologic Cancer
Keywords: Malignant neoplasms of female genital organs; Open gynecologic surgery; Local wound infiltration; Gynecologic cancer; Bupivacaine; Liposomal Bupivacaine; Oxycodone; ETH-Oxydose [DSC]; OxyContin; OxyIR; Roxicodone; Questionnaires; Surveys; MD Anderson Symptom Inventory; MDASI; Pill diary; Medication log
MeSH Terms: interventions — Bupivacaine; Oxycodone; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Group (Active Comparator): Local wound infiltration with Bupivacaine immediately prior to wound closure during gynecological surgery.
  Participants discharged with analgesic opioid regimen of Oxycodone 1-2 tabs (5 mg) by mouth every 4 hours as needed for pain.
  Participants complete a pill diary every day for 30 days after hospital discharge.
  Participants called or emailed and asked questions about symptoms three (3) and 7 days after hospital discharge, and then 1 time every week after that for a total of 8 weeks.
  Interventions: Drug: Bupivacaine; Drug: Oxycodone; Behavioral: Pill Diary; Behavioral: Symptom Questionnaire
- Liposomal Bupivacaine + Bupivacaine Group (Experimental): Local wound infiltration with Liposomal Bupivacaine and 0.25% Bupivacaine admixed immediately prior to wound closure during gynecological surgery.
  Participants discharged with analgesic opioid regimen of Oxycodone 1-2 tabs (5 mg) by mouth every 4 hours as needed for pain.
  Participants complete a pill diary every day for 30 days after hospital discharge.
  Participants called or emailed and asked questions about symptoms three (3) and 7 days after hospital discharge, and then 1 time every week after that for a total of 8 weeks.
  Interventions: Drug: Bupivacaine; Drug: Liposomal Bupivacaine; Drug: Oxycodone; Behavioral: Pill Diary; Behavioral: Symptom Questionnaire

INTERVENTIONS:
Drug: Bupivacaine — 150 mg (0.25%) injected on each side of the wound at the end of surgery before wound closure.
Drug: Liposomal Bupivacaine — 266 mg injected on each side of the wound at the end of surgery before wound closure.
  Arms: Liposomal Bupivacaine + Bupivacaine Group
Drug: Oxycodone — 1-2 tabs (5 mg) by mouth every 4 hours as needed for pain.
  Other Names: ETH-Oxydose [DSC]; OxyContin; OxyIR; Roxicodone
Behavioral: Pill Diary — Participants complete a pill diary every day for 30 days after hospital discharge.
  Other Names: Medication log
Behavioral: Symptom Questionnaire — Participants called or emailed and asked questions about symptoms three (3) and 7 days after hospital discharge, and then 1 time every week after that for a total of 8 weeks.
  Other Names: Survey; MD Anderson Symptom Inventory; MDASI

SUMMARY:
Bupivacaine is a drug that is traditionally given as an injection to numb surgical sites. Liposomes are molecules that are similar to fats. Sometimes drugs are combined with liposomes to make them able to stay in the body for longer periods of time. This has been done with bupivacaine to create liposomal bupivacaine.

The goal of this clinical research study is to compare the effects of bupivacaine to those of liposomal bupivacaine when given to patients who are having gynecologic surgery. Researchers want to compare how long the drugs work to numb the wound and how long patients take to recover from surgery.

DETAILED DESCRIPTION:
Study Arms and Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study arms:

* If you are in Arm 1, you will receive bupivacaine only.
* If you are in Arm 2, you will receive a combination of liposomal bupivacaine and bupivacaine.

You will have an equal (50/50) chance of being assigned to either group. You will not know what you are receiving. However, the study staff will know what you are receiving.

In both cases, the drug(s) will be injected into your skin and tissue at the end of your surgery, right before the wound is closed.

Study Data Collection:

Every day while you are in the hospital recovering from surgery, you will be asked questions about pain, any side effects you may be having, symptoms, and opioid use.

Within 30 days after you leave the hospital, you may also be called and asked about side effects you may be having. If you are called, this call should last about 10-15 minutes. This information may also be collected during a routinely scheduled clinic visit and from the medical record.

Three (3) and 7 days after you leave the hospital, and then 1 time every week after that for a total of 8 weeks, you will be called or emailed and asked questions about any symptoms you may be having. If you are called, each call should last about 10-15 minutes.

If you are also enrolled on the study BS99-094 "Measuring the Symptom Distress of Cancer Patients: Development of a New Assessment System," information from your participation in this study may also be collected and used in that study.

Length of Study:

Your participation on this study will be over 8 weeks after you leave the hospital.

This is an investigational study. Both bupivacaine and liposomal bupivacaine are FDA approved and commercially available. It is investigational to compare the 2 drugs.

Up to 200 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing an exploratory laparotomy for suspected gynecologic cancer, which includes metastatic disease from neoplasia originating in other organs
2. Planned participation in the Gynecologic Enhanced Recovery Pathway
3. Female 18 years of age or older
4. Patient must be able to read and speak English
5. Consents to being part of a randomized, single-blinded study
6. Patient has physical and mental capabilities to take part in study
7. Bilirubin less than or equal to 1.5 x upper limit of the normal range (ULN); Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic-Pyruvic Transaminase (SGPT) </=2.5 x ULN
8. If the patient is of childbearing potential, the patient must have a negative blood or urine pregnancy test within 14 days of surgical treatment on study

Exclusion Criteria:

1. Sensitivity to amide-type local anesthetics
2. Patients on long-acting opioid medications, or scheduled (four or more times a day for seven or more days) short-acting opioid medications within the last 30 days
3. Emergency surgery of any type that does not allow for proper time for protocol review by the patient
4. Surgery that involves known/anticipated resection of anterior abdominal wall with plastic surgery reconstruction
5. Patients undergoing pelvic exenteration
6. Patients undergoing known/anticipated anterior abdominal wall hernia repairs
7. Patients weighing <50 kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Meyer LA, Corzo C, Iniesta MD, Munsell M, Shi Q, Pitcher B, Lasala J, Cain KE, Wang XS, Mena G, Ramirez PT. A prospective randomized trial comparing liposomal bupivacaine vs standard bupivacaine wound infiltration in open gynecologic surgery on an enhanced recovery pathway. Am J Obstet Gynecol. 2021 Jan;224(1):70.e1-70.e11. doi: 10.1016/j.ajog.2020.07.017. Epub 2020 Jul 16. PMID 32682856
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were consented during preoperative visit at MD Anderson Cancer Center from August 31st 2016 to August 31st 2017.
Pre-assignment Details: One patient was excluded after randomization because of scheduled opioid use, and 2 patients were excluded because the surgical approach changed to minimally invasive surgery (these 3 patients were never treated). All patients treated completed the trial.
Groups:
- Active Comparator: Bupivacaine Group: Local wound infiltration with Bupivacaine immediately prior to wound closure during gynecological surgery. Participants discharged with analgesic opioid regimen of Oxycodone 1-2 tabs (5mg) by mouth every 4 hours as needed for pain. Participants complete a pill diary every day for 30 days after hospital discharge. Participants called or emailed and asked questions about symptoms 3 and 7 days after hospital discharge, and then 1 time every week after that for a total of 8 weeks.
- Experimental: Liposomal Bupivacaine + Bupivacaine Group: Local wound infiltration with Liposomal Bupivacaine and 0.25% Bupivacaine admixed immediately prior to wound closure during gynecological surgery. Participants discharged with analgesic opioid regimen of Oxycodone 1-2 tabs (5 mg) by mouth every 4 hours as needed for pain. Participants complete a pill diary every day for 30 days after hospital discharge. Participants called or emailed and asked questions about symptoms 3 and 7 days after hospital discharge, and th3en 1 time every week after that for a total of 8 weeks.
Period: Overall Study
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group
Started | 54 | 48
Completed | 54 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group | Total
Number analyzed (Participants) | 54 | 48 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 37 | 70
  >=65 years | 21 | 11 | 32
Age, Continuous [Median (Full Range); unit: years] | 62.5 [20 to 84] | 59 [22 to 81] | 61 [20 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 37 | 78
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 0 | 6
  White | 40 | 37 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 48 | 102

OUTCOME MEASURES:

1. Primary Outcome: Participants Opioid-Free After Gynecologic Surgery for 48 Hours
Description: Treatment arms compared with respect to the proportion of patients opioid-free at 48 hours using the Cochran-Mantel-Haenszel test stratified by surgeon.
Time Frame: 48 hours
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group
Number analyzed (Participants) | 54 | 48
percentage of participants | 14.8 [6.7 to 27.1] | 16.70 [7.4 to 30.2]

2. Secondary Outcome: Participants Opioid-Free After Gynecologic Surgery
Description: Treatment arms compared with respect to the number of opioid-free days using the Cochran-Mantel-Haenszel test stratified by surgeon.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group
Number analyzed (Participants) | 54 | 48
Participants | 6 | 8

3. Secondary Outcome: Symptom Scores
Description: Daily pain scores were ascertained by routine nursing care every 4 hours while awake, on a 0 to 10 scale. Descriptive statistics and graphical methods used to summarize MD Anderson Symptom Inventory (MDASI) scores at each assessment time by treatment arm. For each symptom component, individuals were asked to rank symptom severity during the previous 24 hours on a scale of 0 to 10, with 0 being "not present "and 10 being "as bad as you can imagine". Symptom interference was also assessed on a 0 to 10 scale, with 0 being "did not interfere" and 10 being "interfered completely". Higher values represent worst outcomes.
Time Frame: Days 0, 2 and 4 postoperatively, up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group
Number analyzed (Participants) | 54 | 48
score on a scale
  Median daily pain scores Postoperative day 0 | 2.5 [1.5 to 4.0] | 2.7 [1.6 to 4.2]
  Median daily pain scores Postoperative day 2 | 2.2 [0.6 to 3.5] | 2.5 [1.0 to 3.0]
  Median daily pain scores Postoperative day 4 | 0.8 [0.2 to 3.0] | 1.2 [0.6 to 3.4]

ADVERSE EVENTS:
Time Frame: within 30 days of the surgery
Arm/Group | Active Comparator: Bupivacaine Group | Experimental: Liposomal Bupivacaine + Bupivacaine Group
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/48
Other Adverse Events (participants affected / at risk) | 0/54 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02740114/Prot_SAP_000.pdf